CLINICAL TRIAL: NCT04244019
Title: Differentiating Radionecrosis From Tumour Progression Using Hybrid FLT-PET/MRI in Patients With Brain Metastases Treated With Stereotactic Radiosurgery.
Brief Title: FLT-PET / MRI Brain Mets
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-6056
Record Dates: First submitted 2020-01-02; First posted 2020-01-28 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Brain Metastases; Radionecrosis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain metastasis (BrM) develops in approximately 40% of cancer patients. Stereotactic radiosurgery (SRS) is a form of radiotherapy that delivers high-dose per fraction to individual lesions that is commonly used to treat BrM.

Radionecrosis (RN) is an adverse event that occurs in approximately 10 - 25% of patients 6 - 24 months after treatment with SRS. Tumour progression may also occur due to local failure of treatment. Radionecrosis and tumour progression share very similar clinical features including vomiting, nausea, and focal neurologic findings.

Radionecrosis and tumour progression also share overlapping imaging characteristics. Due to their similarities, physicians need to perform a surgical resection to diagnose the complication. By using a hybrid FLT-PET/MRI scan, the investigators propose that this combination scan will provide robust data with which to differentiate between radionecrosis and tumour progression without the need for surgery. The investigators plan to conduct a single center feasibility study to investigate the potential in differentiating between SRS and tumour progression in patients, including those who may have previously undergone SRS for BrM, who are suspected to have either RN or tumour progression using hybrid FLT-PET/MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Previously treated with SRS for BrM
3. New intracranial lesion with clinical and radiographic findings suspicious for either RN or tumour progression
4. May be planned surgical resection of the lesion in question. The determination that the lesion is appropriate for and may require surgical resection will be made by the multi-disciplinary brain metastasis team. Surgery is preferred but not required. If a patient is planned for surgery, the date does not need to be established and the patient does not need to have consented in order to be eligible for this study, however the imaging procedure will need to occur prior to the date of surgery.
5. A negative serum pregnancy test within the two-week interval immediately prior to PET-MRI imaging for women of child-bearing age
6. Ability to provide written informed concern to participate in the study

Exclusion Criteria:

1. Previous radiotherapy to the intended treatment volume
2. Active malignancy other than sarcoma
3. Inability to remain supine for at least 60 minutes
4. Pregnancy or breast feeding
5. Age <18 years
6. Failure to provide written informed consent
7. Contraindication for MRI as per current institutional guidelines

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting after being treated with SRS with a new intracranial lesion with clinical and radiographic findings suspicious for either radionecrosis or tumour progression.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Radionecrosis (in patients who have previously received SRS Treatment for BrM) | 24 Months
  Radionecrosis will be assessed by analyzing hybrid FLT-PET/MRI images.

SECONDARY OUTCOMES:
Tumour Progression (in patients who have previously received SRS Treatment for BrM) | 24 Months
  Tumour progression will be assessed by analyzing hybrid FLT-PET/MRI images.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada